CLINICAL TRIAL: NCT06381219
Title: Pediatric Eosinophilic Esophagitis (pedEoE): Effect of Allergen Heat Denaturation on EoE Remission: a Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, Clinic Head in Pediatrics-Allergy at UZ Leuven, Head of the Allergy and Clinical Immunology Research group at KU Leuven (prof., dr.), Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: s67001
Record Dates: First submitted 2023-12-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cow's milk allergen heat denaturation (Other): Children with an EoE in remission AND a previous diet excluding any form of cow's milk will undergo an oral food challenge with extensively heated cow's milk (20'). Afterwards they will be instructed to ensure regular intake of 20' heated cow's milk. After 8 weeks of (re)introduction they will be assessed for potential remaining remission (<15 eosinophils/hpf on esophagal biopsies). If remission is sustained, they will sequentially decrease the degree of heat denaturation by decreasing the cooking time: 15', 10' and 5' cooked cow's milk. At the end, parents will have the choice to add a final step of raw cow's milk. After every 8 weeks of every new step, a gastroscopy will be performed to assess maintained remission. If remission is lost, they will go back to a strict avoidance diet for at least 10 weeks.
  Interventions: Other: Implementation of cow's milk in decreasingly heated forms
- Hen's egg allergen heat denaturation (Other): Children with an EoE in remission AND a previous diet excluding any form of hen's egg will undergo an oral food challenge with strongly heated hen's egg (in cake). Afterwards they will be instructed to ensure regular intake of cake. After 8 weeks of (re)introduction they will be assessed for potential remaining remission (<15 eosinophils/hpf on esophagal biopsies). If remission is sustained, they will sequentially decrease the degree of heat denaturation as follows: hard-boiled egg, omelet and soft-boiled egg. At the end, parents will have the choice to add a final step of raw egg. After every 8 weeks of every new step, a gastroscopy will be performed to assess maintained remission. If remission is lost, they will go back to a strict avoidance diet for at least 10 weeks.
  Interventions: Other: Implementation of hen's egg in decreasingly heated forms

INTERVENTIONS:
Other: Implementation of cow's milk in decreasingly heated forms — Implementation of cow's milk in decreasingly heated forms to assess maintained remission of EoE
  Arms: Cow's milk allergen heat denaturation
Other: Implementation of hen's egg in decreasingly heated forms — Implementation of hen's egg in decreasingly heated forms to assess maintained remission of EoE
  Arms: Hen's egg allergen heat denaturation

SUMMARY:
The objective of the study is to study whether the introduction of heated food products (more specifically heated hen's egg and/or cow's milk) in children with EoE would be possible without re-occurrence of the eosinophilic inflammation, while the intake of less heated products might cause disease recidive. Moreover, we would like to study whether the gradual re-introduction of less heated products after the most heated form is tolerated, could lead to tolerance induction in EoE.

DETAILED DESCRIPTION:
If inclusion criteria are met, after obtaining informed consent from the parents (and when old enough, assent from the children) children with cow's milk and/or hen's egg induced pedEoE will be included in this pilot trial. Baseline blood will be obtained before in-house OFC procedure and serum will be stored for specific IgG4 analysis. In parallel, PBMCs will be isolated and stimulated in vitro with heat denatured proteins. B cells will be stained by 4-laserflow cytometry. IgG4 production in supernatants will be studied by ELISA (specific IgG4 by Immunocap 100). This procedure will be repeated during each gastroscopy.

Children will be provoked in-house, based on the written procedure available for heated egg or cow's milk provocation. Afterwards, they will introduce heated egg by cake or 20' boiled cow's milk at least three times a week for 8 weeks and will return to the hospital for a gastroscopy with biopsies. EoE remission will be studied on biopsies of the upper and lower esophagus by eosinophil staining within the routine anatomopathological laboratory within our hospital.

If remission remains, subjects will be invited to introduce less heated hen's egg or cow's milk for 8 weeks, after which they will return to the hospital for the second gastroscopy with similar procedure. This is repeated three times until 4' soft-boiled egg or 5' boiled cow's milk is introduced for 8 weeks. When remission remains after this introduction, the children and parents are offered the possibility to terminate the study or to introduce either raw egg (tiramisu or chocolate mousse) or uncooked UHT-treated cow's milk for 8 weeks after which gastroscopy with biopsies will be performed.

If remission is lost, they will return to the strict avoidance diet for at least 10 weeks after which they will return to the hospital for their second gastroscopy. Upon remission after avoidance, the children will remain eligible for another heat denatured food challenge (when on diet for both).

ELIGIBILITY:
Inclusion Criteria:

All children (aged 12 months and older) presenting (since 1-1-2014: moment of diagnostic guideline standardization for pedEoE) with diagnosed pedEoE at UZ Leuven eliminating either hen's egg or cow's milk or both and in complete remission after their latest biopsy (no longer than 12 months earlier, but preferentially as short as possible after their latest biopsy) are eligible for the study. If the last biopsy has been performed more than 12 months earlier, a new gastro-duodenoscopy will be performed to verify remission and rule out e.g. active gastritis. If they are on PPI and/or local budesonide treatment, this should be stable for at least 3 months and will remain untouched during the entire study. We will include 18 pedEoE subjects suffering from cow's milk induced EoE and 18 suffering from hen's egg induced EoE.

Exclusion Criteria:

* Children younger than 12 months
* Children with active pedEoE
* Children who refuse to adhere to the protocol
* Children with associated IgE mediated hen's egg and/or cow's milk allergy with specific IgE antibody titers that predict active (baked egg and/or baked milk) food allergy with cut-off titers as used at the consultation of allergy (KLL). Those children will become eligible however if their titers decrease while the study is still open.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maintained remission of EoE | 40 weeks
  Primary end-point of the study is to study the number of pedEoE children by inclusion on hen's egg and/or cow's milk free diet with potential remaining remission (<15 eosinophils/hpf on esophageal biopsies) after 8 weeks (re)introduction of heat-denatured hen's egg and/or cow's milk proteins (introduced sequentially as on the one hand baked egg (cake), hard-boiled egg, omelet and soft-boiled egg and on the other hand 20' cooked cow's milk, 15', 10' and 5' cooked cow's milk).

SECONDARY OUTCOMES:
Maintained remission only in step 1 of the diet | Assessment of failed remission 8 weeks after step 2 but successful remission after step 1
  The number of pedEoE children in whom remission remain with introduction of cake and/or 20' cooked cow's milk (step 1), but no longer with less heated proteins.
Association of remission with circulating IgG4 levels | Bloods will be taken during every gastroscopy
  To study whether remission (>15 eosinophils per high-power field) is associated with specific circulating and/or local food protein IgG4 reduction (and increase upon unsuccessful introduction of less heated proteins). We will compare the IgG4 levels (expressed in g/L) in patients in remission and those not in remission.
Association of remission with IgG4 levels on biopsy | At every gastroscopy
  To study whether remission (>15 eosinophils per high-power field) can be associated with changes in local IgG4 production that will be measured by biopsy staining and expressed in number of IgG4 positive plasma cells per high-power field. We will compare the local IgG4 production in patients in remission and those not in remission.
In vitro B cell test to mimic B cell activation after stimulation | Up to 6 months
  After PBMC isolation from the blood of pediatric patients, the PBMCs will be in vitro stimulated with food proteins. Then, B cell activation will be measured with flow cytometry by looking at the proportion of activated B cells compared to the total number of B cells.
Correlation between QoL and remission | Up to 45 weeks
  Can we observe a correlation between Pediatric EoE PEESS v2.0 and Peds-QL scores (obtained in all pedEoE children participating in study s64441) and histologic remission?
Associated atopy | On inclusion with initial characteristics of the patients
  To study the presence of associated atopy (tree-, grass- or weed pollen or fungi allergy).
Associated food allergies | On inclusion with initial characteristics of the patients
  To study the presence of associated typical IgE mediated food allergy (sensitization and documented symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Hoffman, Prof. Dr., Principal Investigator — Co-investigator, pediatric gastro-enterology; Gert De Hertogh, Prof. Dr., Principal Investigator — Co-investigator, pathological anatomy
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

DOCUMENTS (1):
  • Study Protocol (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06381219/Prot_000.pdf